CLINICAL TRIAL: NCT05326776
Title: Effect of Peripheral Oxytocin on Touch Pleasantness and Pain
Brief Title: Peripheral Oxytocin and Touch
Acronym: POPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Laura Case, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 802467
Record Dates: First submitted 2022-04-04; First posted 2022-04-14 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Order 1 (Experimental): Participants will receive 4mcg/2ml oxytocin during Session 1 and 2ml isotonic saline during Session 2, injected into the forearm.
  Interventions: Drug: Pitocin
- Order 2 (Experimental): Participants will receive 2ml isotonic saline during Session 1 and 4mcg/2ml oxytocin during Session 2, injected into the forearm.
  Interventions: Drug: Pitocin

INTERVENTIONS:
Drug: Pitocin — At each session, 4mcg/2ml oxytocin or 2ml isotonic saline (0.9% sodium chloride; placebo control) will be injected into the middle of the dorsal forearm. Sessions will be separated by at least 48 hours to ensure drug clearance.

SUMMARY:
Research shows that slow gentle skin stroking can activate special sensory nerves in the skin that elicit relaxing effects on the body and mind, similar to the effects of the hormone oxytocin. Studies also suggest that gentle stroking may even release oxytocin in the skin. However, we do not know what oxytocin does in the skin and how it affects nerves that send pleasant touch or pain signals to the brain. The proposed study will determine how individuals perceive gentle stroking and experimental pain before and after a skin injection of oxytocin compared to a placebo injection.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 65 years old
2. Fluent in English
3. Healthy

   Exclusion Criteria:
4. Sensory or motor nerve deficit
5. Acute or chronic pain
6. Major medical conditions such as kidney, liver, cardiovascular (hypertension, preexisting cardiac arrhythmia), autonomic, pulmonary, or neurological problems (e.g., seizure disorder) or a chronic systemic disease (e.g., diabetes).
7. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
8. Unstable psychiatric conditions
9. Needle phobia or history of fainting
10. Current use of opiate medication(s)
11. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
12. Currently pregnant or pregnant within the last two years
13. Currently nursing or lactating
14. Current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval
15. Past or current history of hyponatremia or at risk for hyponatremia
16. Current use of thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, Ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, selective serotonin reuptake inhibitors, monoamine oxidase inhibitora, or the recreational drug ecstasy
17. Latex allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ACTRI, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared with other researchers per request.
Supporting Information: Study Protocol
Time Frame: Upon study completion for as long as possible.
Access Criteria: For academic researchers conducting reviews, meta-analyses, or secondary analyses.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited from the local community as well as from our previous studies. Potential participants completed a telephone screening during which the study procedures were described, and eligibility criteria were reviewed.
Pre-assignment Details: Screening was conducted prior to enrollment. No participants were excluded after enrollment.
Period: Overall Study
Arm/Group | Order 1 | Order 2
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Order 1 | Order 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (12.5) | 26.2 (6.5) | 27.4 (9.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  gender: female | 5 | 7 | 12
  gender: non-binary | 1 | 0 | 1
  gender: male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Pleasantness Rating of Gentle Brushing
Description: Touch pleasant/unpleasantness ratings will be assessed in response to slow gentle brushing using a "Pleasantness/Unpleasantness" Visual Analog Scale with anchors of "Extremely unpleasant" (coded -100) to "Neutral" to "Extremely pleasant (coded 100)." Change in mean rating of slow brushing will be compared between the oxytocin and placebo sessions. Higher values indicate increased pleasantness (better outcome).
Time Frame: Baseline and time of intervention at both the Oxytocin Session and Placebo Session (Sessions spaced a minimum of 3 days apart)
Population: All participants who completed both sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Oxytocin Session: Data from during the Oxytocin Session, regardless of order.
- Placebo Session: Data from during the Placebo saline Session, regardless of order.
Arm/Group | Oxytocin Session | Placebo Session
Number analyzed (Participants) | 18 | 18
score on a scale | -8.7 (23.0) | -14.1 (27.8)

2. Primary Outcome: Change in Mechanical Threshold
Description: "Mechanical threshold" task. Change in first reported percept of sharpness from application of a standard set of weighted pinprick stimuli (minimum 8mN; maximum 512 mN) will be compared between the oxytocin and placebo sessions. An increased threshold indicates reduced sensitivity to mechanical pain.
Time Frame: as for outcome 1
Population: All participants who completed both sessions.
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | Oxytocin Session | Placebo Session
Number analyzed (Participants) | 18 | 18
mN | 65.3 (143.1) | 63.2 (125.9)

3. Primary Outcome: Change in Temporal Summation of Pinprick Stimuli
Description: Temporal summation will be tested using a standard 256 milliNewtons (mN) pinprick stimulus applied for 10 repetitions. The participant will provide pain ratings for a single pinprick and for the 10 repetitions, using a Visual Analog Scale rating scale with anchors "No pain" to "Most intense pain imaginable." This procedure will be repeated 5 times and the mean pain rating for the repeated pinprick will be divided by the mean rating of the single pinprick to obtain the standard temporal summation ratio. Change in ratio will be compared between the oxytocin and placebo sessions.
Time Frame: as for outcome 1
Population: All participants who completed both sessions.
Measure: Mean (Standard Deviation); unit: change in ratio of ratings on scales
Arm/Group | Oxytocin Session | Placebo Session
Number analyzed (Participants) | 18 | 18
change in ratio of ratings on scales | 0.15 (0.63) | -.02 (1.3)

4. Secondary Outcome: Pressure Pain Threshold
Description: Pressure pain threshold will be tested using a pressure algometer placed over the dorsal forearm muscles, and pressure will be increased until pain is reported. When pain is reported, the pressure level (in pounds of force) is recorded as the outcome measure.
Time Frame: as for outcome 1
Population: All participants who completed both sessions.
Measure: Mean (Standard Deviation); unit: changes in pounds of force
Arm/Group | Oxytocin Session | Placebo Session
Number analyzed (Participants) | 18 | 18
changes in pounds of force | 0.13 (1.9) | 0.58 (1.5)

5. Secondary Outcome: Heat Pain Threshold
Description: Heat pain threshold (HPT) will be tested using a high-quality thermode. To establish HPT, the thermode will be placed on the arm at a baseline temperature of 32 Celsius and will be increased until the stimulus is reported as painful by the participant. The mean of three trials will be taken as the HPT.
Time Frame: as for outcome 1
Population: All participants who completed both sessions.
Measure: Mean (Standard Deviation); unit: changes in degrees Celsius
Arm/Group | Oxytocin Session | Placebo Session
Number analyzed (Participants) | 18 | 18
changes in degrees Celsius | 0.3 (2.5) | -0.29 (1.3)

6. Secondary Outcome: Heat Pain Ratings
Description: Three 10s trials of the individually calibrated heat stimulus rated 70/100 will be rated using using a "Pain Intensity" Visual Analog Scale rating scale with anchors "No pain" (coded -100) to "Most intense pain imaginable (coded 100)." Higher scores indicate more intense pain (worse outcome).
Time Frame: as for outcome 1
Population: All participants who completed both sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin Session | Placebo Session
Number analyzed (Participants) | 18 | 18
score on a scale | -15.0 (43.9) | 1.2 (23.5)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Groups:
- Oxytocin Session: Data from during the Oxytocin Session, regardless of order.
  4mcg/2ml oxytocin was injected into the middle of the dorsal forearm.
- Placebo Session: Data from during the Placebo Session, regardless of order.
  2ml isotonic saline was injected into the forearm.
Arm/Group | Oxytocin Session | Placebo Session
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT05326776/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT05326776/ICF_001.pdf